CLINICAL TRIAL: NCT06449391
Title: A Clinical Exploratory Study of Root Analogy Implant
Brief Title: The Application of Root Analogy Implant in Immediate Implantation
Acronym: RAI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024035
Record Dates: First submitted 2024-05-27; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Dental Implantation; Dental Implants; Osseointegration
Keywords: root analogy implant; Immediate implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- implanted group (Experimental): This study is a single arm study, with only immediate implantation of root analogy implants
  Interventions: Device: RAI

INTERVENTIONS:
Device: RAI — Immediate implantation

SUMMARY:
The current clinical implant techniques used include immediate implantation, early implantation, and delayed implantation. With the acceleration of the current pace of life, immediate implantation is increasingly favored by patients due to its advantages such as fewer surgeries, shorter waiting times, and less impact on aesthetics. The research group has shown that the mismatch between traditional implants and extraction sockets in immediate implantation surgery has caused some complications. Therefore, it is believed that 3D printed personalized root shaped implants with certain roughness are more suitable for use in immediate implantation surgery.

DETAILED DESCRIPTION:
The current clinical implant techniques used include immediate implantation, early implantation, and delayed implantation. With the acceleration of the current pace of life, immediate implantation is increasingly favored by patients due to its advantages such as fewer surgeries, shorter waiting times, and less impact on aesthetics. The research group has shown that the mismatch between traditional implants and extraction sockets in immediate implantation surgery has caused some complications. Therefore, it is believed that 3D printed personalized root shaped implants with certain roughness are more suitable for use in immediate implantation surgery. A 3D printed personalized root implant system jointly developed by Zhejiang University School of Medicine Affiliated Stomatology Hospital, Zhejiang University School of Mechanical Engineering, and Hangzhou Ya Natural Technology Co., Ltd. The implant part of this implant system is implanted into the bone using laser melting printing technology in additive manufacturing methods. The raw material is pure titanium powder, and research results in New Zealand white rabbits and beagles have confirmed that the implant has good bone bonding ability, which can shorten surgical time, reduce surgical frequency, compress implant cycle, restore chewing function, and other advantages. The relevant research results have been published in the top oral journal Journal of Dental Research, and the chemical composition and biological safety of the material have been tested by the Zhejiang Medical Device Inspection and Research Institute (test report number: Z20221903), Z20222527，G20233158）。 The base and other accessories are cut from titanium rods using conventional reduction manufacturing techniques.

ELIGIBILITY:
Inclusion Criteria:

* Age:20-60 years old, gender unlimited
* Good oral hygiene
* No systemic diseases
* There are irreparable residual roots, no obvious apical periodontitis, no looseness greater than degree II, and the tooth position includes four quadrant anterior teeth and premolars
* Root length greater than 10 mm, and no significant bone resorption at the alveolar crest
* There is no significant displacement of adjacent teeth and no significant elongation of opposing teeth
* The bone density of the target implant area is Class II and Class III
* The lateral bone wall of the lips (cheeks), palate (tongue) is intact and larger than 1mm
* The subjects are able to understand the purpose of the experiment, willing to -cooperate with surgical treatment and follow-up, voluntarily participate in the experiment, and sign an informed consent form.

Exclusion Criteria:

* Patients with moderate to severe periodontitis
* Missing proximal and distal adjacent teeth in the target residual root
* Residual roots with root adhesion
* The target implant area has a bone density of Class I or IV
* Acute infectious disease or metabolic bone disease activity period
* Patients with diabetes history and poor blood glucose control (fasting blood glucose ≥ 8.8 mmol/L L)
* Patients with liver and kidney dysfunction (AST, ALT ≥ 1.5 times ULNULN, creatinine ≥ 1.5 times ULNULN)
* Individuals with a history of osteoporosis
* Individuals with a history of malignant tumors or other serious illnesses who are not suitable for surgery
* Individuals with mental disorders and lack of autonomous behavior ability Pregnant women, lactating or menstruating women, and women with pregnancy plans within six months
* Various possible causes of imaging artifacts in the surgical area
* Receiving medication that may affect bone metabolism (such as bisphosphonates) within the past 3 months
* The researchers estimate poor compliance or other factors that are not suitable for conducting this experiment.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Alveolar ridge height | day 0,12 weeks,24weeks,48weeks
  The distance from the top of the alveolar ridge to the tip of the implant

SECONDARY OUTCOMES:
Width of alveolar ridge, buccal and lingual directions | day 0，12 weeks, 24 weeks, 48 weeks
  The width of the implant platform from the buccal and lingual to the alveolar bone
Implant mobility | day 0，12 weeks
  Measure the movement of the implant using an implant mobility meter and record the ISQ value
Gingival condition | day 0, 12 weeks, 24 weeks, 48weeks
  Two independent clinical doctors conducted gingival examination in the oral implant area of the patient, and gave a comprehensive score for gingival condition based on changes in gingival color, shape, and texture. A 3-point scoring method was used, with good, average, and poor results.
Exploration depth and Exploring bleeding | 12 weeks, 24 weeks, 48 weeks
  Same periodontal probing. Use blunt head periodontal probing to measure the depth of probing at six points around the implant, including the buccal mesial, buccal central, buccal distal, lingual palatal mesial, lingual palatal central, and lingual palatal distal. Record the depth of probing and calculate the average value, 2-4mm if normal, if depth >5mm, consider the occurrence of periimplantitis. The improved gingival sulcus bleeding index (mSBI) can be used to detect bleeding: 0=Along the periphery of the implant, no bleeding after soft tissue edge exploration; 1=scattered points after exploration, hemorrhage in shape; 2=After diagnosis, the bleeding appears linear in the groove; 3=severe or Spontaneous bleeding.
Clinical looseness of implants | 12 weeks, 24 weeks, 48 weeks
  Evaluation of tooth looseness. Use tweezers to clamp and shake the cutting edge during the examination of anterior dental implants; When checking the posterior dental implant, fold the forceps together and place them in the center of the occlusal fissure, shaking them towards the buccal, lingual (palatal), and mesial and distal directions (clamping the anterior tooth ridge, and pressing the posterior tooth forceps against the posterior occlusal fissure). The commonly used method for recording tooth looseness in clinical practice is to calculate the degree of looseness in millimeters: degree I looseness: the looseness amplitude is within 1mm; Second degree loosening: the loosening amplitude is within 1-2mm; Third degree loosening: the loosening amplitude is above 2mm.
Recovery of chewing function | 24 weeks, 48 weeks
  The basic method is to use a vernier ruler about 10 cm long, where "0" represents complete dissatisfaction and "10" represents complete satisfaction. The patient marks the line segment based on their own satisfaction, and the physician scores them based on the position marked by the patient.
Aesthetic satisfaction | 24 weeks，48 weeks
  Use a survey questionnaire to evaluate patient satisfaction, including aesthetics and other suggestions and opinions on treatment. The evaluation adopts a 3-point scoring method, which is satisfied, average, and dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Stomatology Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China